CLINICAL TRIAL: NCT00454636
Title: Open Label, Phase II Study of Capecitabine (Xeloda®) as Fluoropyrimidine of Choice in Combination With Chemotherapy in Patients With Advanced and/or Metastatic Gastric Cancer Suitable for Treatment With a Fluoropyrimidine-Based Regimen
Brief Title: A Study of Xeloda (Capecitabine) in Combination With Chemotherapy in Patients With Advanced and/or Metastatic Gastric Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20777
Record Dates: First submitted 2007-03-30; First posted 2007-04-02 (Estimated); Results first posted 2016-08-19 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; Capecitabine; Epirubicin; Oxaliplatin; Docetaxel

ARMS (4):
- Cisplatin / Capecitabine (Experimental): Cisplatin, 80 mg/m2/day, intravenous (IV), every 3 weeks; capecitabine, 1,000 mg/m2, oral, twice daily for 2 weeks, followed by 1 week of rest in each cycle. Study drugs were administered for at least 24 weeks.
  Interventions: Drug: Cisplatin; Drug: Capecitabine
- Epirubicin / Cisplatin / Capecitabine (Experimental): Epirubicin, 50 mg/m2/day, IV, every 3 weeks; cisplatin, 60 mg/m2/day, IV, every 3 weeks; capecitabine, 625mg/m2, orally, twice daily per 3-week cycle. Study drugs were administered for at least 24 weeks.
  Interventions: Drug: Epirubicin; Drug: Cisplatin; Drug: Capecitabine
- Epirubicin / Oxaliplatin / Capecitabine (Experimental): Epirubicin, 50 mg/m2/day, IV, every 3 weeks; oxaliplatin, 130 mg/m2/day, IV, every 3 weeks; capecitabine, 625mg/m2 orally, twice daily per 3-week cycle. Study drugs were administered for at least 24 weeks.
  Interventions: Drug: Epirubicin; Drug: Capecitabine; Drug: Oxaliplatin
- Docetaxel / Cisplatin / Capecitabine (Experimental): Docetaxel, 60 mg/m2/day, IV, every 3 weeks; cisplatin, 60 mg/m2/day, IV, every 3 weeks; capecitabine, 825 mg/m2, orally, twice daily for 2 weeks, followed by 1 week of rest in each cycle. Study drugs were administered for at least 24 weeks.
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Drug: Capecitabine

INTERVENTIONS:
Drug: Cisplatin — 80 mg/m2/day, intravenous (IV), every 3 weeks
  Arms: Cisplatin / Capecitabine
Drug: Capecitabine — 1,000 mg/m2, oral, twice daily for 2 weeks, followed by 1 week of rest in each cycle
  Other Names: Xeloda
  Arms: Cisplatin / Capecitabine
Drug: Epirubicin — 50 mg/m2/day, IV, every 3 weeks
  Arms: Epirubicin / Cisplatin / Capecitabine; Epirubicin / Oxaliplatin / Capecitabine
Drug: Cisplatin — 60 mg/m2/day, IV, every 3 weeks
  Arms: Docetaxel / Cisplatin / Capecitabine; Epirubicin / Cisplatin / Capecitabine
Drug: Capecitabine — 625 mg/m2, oral, twice daily per 3-week cycle
  Other Names: Xeloda
  Arms: Epirubicin / Cisplatin / Capecitabine; Epirubicin / Oxaliplatin / Capecitabine
Drug: Oxaliplatin — 130 mg/m2/day, IV, every 3 weeks
  Arms: Epirubicin / Oxaliplatin / Capecitabine
Drug: Docetaxel — 60 mg/m2/day, IV, every 3 weeks
  Arms: Docetaxel / Cisplatin / Capecitabine
Drug: Capecitabine — 825 mg/m2, oral, twice daily for 2 weeks
  Other Names: Xeloda
  Arms: Docetaxel / Cisplatin / Capecitabine

SUMMARY:
This study will assess the safety and efficacy of Xeloda, given in combination with standard chemotherapy regimens, for the first-line treatment of advanced and/or metastatic gastric cancer. All patients will receive Xeloda in combination with one of 4 standard chemotherapy regimens; the dose of Xeloda will be from 625mg/m2 - 1000mg/m2 bid orally, depending on the chemotherapy regimen used. The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* advanced or metastatic gastric cancer;
* Eastern Cooperative Oncology Group (ECOG) <=2.

Exclusion Criteria:

* previous chemotherapy (except adjuvant or neoadjuvant treatment >=6 months prior to study);
* evidence of central nervous system (CNS) metastasis;
* history of another malignancy within the last 5 years (except for successfully treated basal cell cancer of skin, or in situ cancer of the cervix);
* clinically significant cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2007-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (41):
- Spain (41):
  - Alcoy, Alicante
  - Ávila, Avila
  - Palma de Mallorca, Balearic Islands
  - Barcelona, Barcelona
  - Burgos, Burgos
  - Cadiz, Cadiz
  - Jerez de la Frontera, Cadiz
  - Puerto Real, Cadiz
  - Castellon, Castellon
  - Córdoba, Cordoba
  - Girona, Girona
  - Granada, Granada
  - Guadalajara, Guadalajara
  - Donostia / San Sebastian, Guipuzcoa
  - Barbastro, Huesca
  - Huesca, Huesca
  - Jaén, Jaen
  - A Coruña, La Coruña
  - Ferrol, La Coruña
  - Santiago de Compostela, La Coruña
  - Logroño, La Rioja
  - León, Leon
  - Lleida, Lerida
  - Lugo, Lugo
  - Alcorcón, Madrid
  - Madrid, Madrid
  - Murcia, Murcia
  - Navarra, Navarre
  - Pamplona, Navarre
  - Ourense, Orense
  - Palencia, Palencia
  - Pontevedra, Pontevedra
  - Vigo, Pontevedra
  - Gijón, Principality of Asturias
  - Salamanca, Salamanca
  - Seville, Sevilla
  - San Cristóbal de La Laguna, Tenerife
  - Toledo, Toledo
  - Valencia, Valencia
  - Bilbao, Vizcaya
  - Zaragoza, Zaragoza

RESULTS

PARTICIPANT FLOW:
Groups:
- Cisplatin / Capecitabine: Cisplatin, 80 mg/m2/day, intravenous (IV), every 3 weeks; capecitabine, 1,000 mg/m2, orally, twice daily for 2 weeks, followed by 1 week of rest in each cycle. Study drugs were administered for at least 24 weeks
Period: Overall Study
Arm/Group | Cisplatin / Capecitabine | Epirubicin / Cisplatin / Capecitabine | Epirubicin / Oxaliplatin / Capecitabine | Docetaxel / Cisplatin / Capecitabine
Started | 41 | 32 | 27 | 58
Completed | 10 | 9 | 7 | 26
Not Completed | 31 | 23 | 20 | 32
Not completed — Adverse Event | 10 | 6 | 9 | 15
Not completed — Disease Progression | 11 | 12 | 4 | 11
Not completed — Protocol Violation | 3 | 2 | 3 | 3
Not completed — Death | 6 | 1 | 1 | 1
Not completed — Patient refusal | 1 | 1 | 3 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cisplatin / Capecitabine | Epirubicin / Cisplatin / Capecitabine | Epirubicin / Oxaliplatin / Capecitabine | Docetaxel / Cisplatin / Capecitabine | Total
Number analyzed (Participants) | 41 | 32 | 27 | 58 | 158
Age, Continuous [Median (Full Range); unit: years] | 66 [39 to 77] | 60 [38 to 78] | 62 [40 to 79] | 58 [20 to 78] | 61 [20 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 9 | 4 | 15 | 46
  Male | 23 | 23 | 23 | 43 | 112

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade 3 Hand-Foot Syndrome (HFS)
Time Frame: Approximately 3.25 years
Population: Safety population: All participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Cisplatin / Capecitabine | Epirubicin / Cisplatin / Capecitabine | Epirubicin / Oxaliplatin / Capecitabine | Docetaxel / Cisplatin / Capecitabine
Number analyzed (Participants) | 41 | 32 | 27 | 58
percentage of participants | 2.4 | 6.3 | 3.7 | 5.2

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants achieving either a complete response (CR) or a partial response (PR), based on Response Evaluation Criteria in Solid Tumors (RECIST) v.1.0 criteria. CR was defined as the disappearance of all target lesions; for non-target lesions, disappearance of lesions and normal tumor marker levels. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, using the baseline sum LD as reference.
Time Frame: Approximately 3.25 years
Population: Intent-to-Treat (ITT) population: included all participants who received at least one dose of study medication and had baseline and at least one subsequent tumor assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cisplatin / Capecitabine | Epirubicin / Cisplatin / Capecitabine | Epirubicin / Oxaliplatin / Capecitabine | Docetaxel / Cisplatin / Capecitabine
Number analyzed (Participants) | 30 | 27 | 23 | 52
percentage of participants | 43.3 [25.5 to 62.6] | 40.7 [22.4 to 61.2] | 69.6 [47.1 to 86.8] | 59.6 [45.1 to 73.0]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the start of treatment to the first documentation of disease progression or death for any cause. Disease progression was based on Response Evaluation Criteria in Solid Tumors (RECIST) v.1.0 criteria and was defined as at least a 20% increase in the sum of LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Approximately 3.25 years
Population: Safety population: All participants who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin / Capecitabine | Epirubicin / Cisplatin / Capecitabine | Epirubicin / Oxaliplatin / Capecitabine | Docetaxel / Cisplatin / Capecitabine
Number analyzed (Participants) | 41 | 32 | 27 | 58
months | 4.43 [3.10 to 7.70] | 5.17 [2.97 to 6.23] | 7.07 [3.03 to 11.23] | 7.87 [5.53 to 9.80]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time elapsing from the date of the start of treatment until death, or last known follow-up.
Time Frame: Approximately 3.25 years
Population: Safety population: All participants who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin / Capecitabine | Epirubicin / Cisplatin / Capecitabine | Epirubicin / Oxaliplatin / Capecitabine | Docetaxel / Cisplatin / Capecitabine
Number analyzed (Participants) | 41 | 32 | 27 | 58
months | 10.23 [4.73 to 12.60] | 8.87 [5.30 to 14.57] | 13.87 [5.37 to 24.07] | 12.43 [10.60 to 15.67]

5. Secondary Outcome: Duration of Response
Description: Duration of Response was defined as the time of complete response (CR) or partial response (PR) until the first date of recurrent or progressive disease, based on Response Evaluation Criteria in Solid Tumors (RECIST) v.1.0 criteria. CR was defined as the disappearance of all target lesions; for non-target lesions, disappearance of lesions and normal tumor marker levels. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, using the baseline sum LD as reference. Progressive disease was defined as at least a 20% increase in the sum of LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Approximately 3.25 years
Population: Safety population: All participants who received at least one dose of study medication. Only participants who reported either a complete response or a partial response were assessed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cisplatin / Capecitabine | Epirubicin / Cisplatin / Capecitabine | Epirubicin / Oxaliplatin / Capecitabine | Docetaxel / Cisplatin / Capecitabine
Number analyzed (Participants) | 13 | 11 | 16 | 31
days | 308.92 (348.44) | 154.09 (167.83) | 203.06 (232.54) | 205.52 (228.44)

6. Secondary Outcome: Time to Response
Description: Time to Response was defined as the date of start of treatment until the first date of complete response (CR) or a partial response (PR), based on Response Evaluation Criteria in Solid Tumors (RECIST) v.1.0 criteria. CR was defined as the disappearance of all target lesions; for non-target lesions, disappearance of lesions and normal tumor marker levels. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, using the baseline sum LD as reference.
Time Frame: Approximately 3.25 years
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cisplatin / Capecitabine | Epirubicin / Cisplatin / Capecitabine | Epirubicin / Oxaliplatin / Capecitabine | Docetaxel / Cisplatin / Capecitabine
Number analyzed (Participants) | 13 | 11 | 16 | 31
days | 132.92 (52.24) | 126.64 (74.69) | 123.50 (60.22) | 138.16 (44.29)

ADVERSE EVENTS:
Time Frame: Approximately 3.25 years
Arm/Group | Cisplatin / Capecitabine | Epirubicin / Cisplatin / Capecitabine | Epirubicin / Oxaliplatin / Capecitabine | Docetaxel / Cisplatin / Capecitabine
Serious Adverse Events (participants affected / at risk) | 9/41 | 12/32 | 12/27 | 23/58
Other Adverse Events (participants affected / at risk) | 39/41 | 30/32 | 27/27 | 54/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin / Capecitabine (N=41) | Epirubicin / Cisplatin / Capecitabine (N=32) | Epirubicin / Oxaliplatin / Capecitabine (N=27) | Docetaxel / Cisplatin / Capecitabine (N=58)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 5
Asthenia (General disorders) | 1 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium (Infections and infestations) | 0 | 0 | 0 | 1
Bacteraemia gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Limb operation (Surgical and medical procedures) | 0 | 1 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin / Capecitabine (N=41) | Epirubicin / Cisplatin / Capecitabine (N=32) | Epirubicin / Oxaliplatin / Capecitabine (N=27) | Docetaxel / Cisplatin / Capecitabine (N=58)
Anaemia (Blood and lymphatic system disorders) | 10 | 12 | 7 | 19
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 4 | 4
Neutropenia (Blood and lymphatic system disorders) | 18 | 10 | 13 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 1 | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 4 | 4
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3 | 2 | 6
Constipation (Gastrointestinal disorders) | 3 | 9 | 6 | 13
Diarrhoea (Gastrointestinal disorders) | 12 | 8 | 13 | 28
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 0 | 7
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 10 | 15 | 10 | 17
Vomiting (Gastrointestinal disorders) | 16 | 17 | 15 | 24
Asthenia (General disorders) | 20 | 14 | 17 | 36
Mucosal inflammation (General disorders) | 7 | 9 | 4 | 11
Oedema (General disorders) | 1 | 0 | 2 | 2
Oedema peripheral (General disorders) | 1 | 3 | 2 | 1
Pain (General disorders) | 2 | 0 | 1 | 3
Pyrexia (General disorders) | 3 | 6 | 3 | 9
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1 | 3
Oral candidiasis (Infections and infestations) | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 3
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 3
Weight decreased (Investigations) | 1 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 9 | 8 | 15
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 4
Dizziness (Nervous system disorders) | 3 | 0 | 5 | 1
Dysaesthesia (Nervous system disorders) | 1 | 0 | 5 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 2 | 3
Neurotoxicity (Nervous system disorders) | 0 | 1 | 3 | 7
Paraesthesia (Nervous system disorders) | 1 | 0 | 6 | 8
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 3
Renal failure (Renal and urinary disorders) | 3 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 15 | 5 | 14
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 9 | 4 | 11
Deep vein thrombosis (Vascular disorders) | 1 | 3 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 2 | 0
Phlebitis (Vascular disorders) | 0 | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.